CLINICAL TRIAL: NCT05288998
Title: Noninvasive Evaluation of the Intrarenal Microvasculature in ADPKD
Brief Title: Intrarenal Microvasculature in ADPKD
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Maria V. Irazabal Mira, Principal Investigator, Mayo Clinic
Other Study IDs: 21-005117; 1R21DK129886-01 (NIH)
Record Dates: First submitted 2022-02-21; First posted 2022-03-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: ADPKD; Intrarenal microvasculature
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and plasma samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with a previous diagnosis of ADPKD: Patients that have been diagnosed with ADPKD and meet the study's inclusion criteria
- Healthy Volunteers: Subjects without a family or personal history of kidney disease or concomitant systemic disorder that might affect the kidney

SUMMARY:
The primary objective of this study is to evaluate the use of Super-resolution ultrasound (SRU) to assess the intrarenal microvasculature in patients with Autosomal Dominant Polycystic Kidney Disease (ADPKD) and healthy volunteers.

DETAILED DESCRIPTION:
An intact intrarenal microcirculation is vital to preserving normal kidney function, and microvascular dysfunction, damage, and loss are known to contribute to renal function decline. In ADPKD, extensive vascular remodeling has been proposed to play an important role in its progression. However, microvascular analyses in rodents and humans with ADPKD have been performed ex vivo or in vitro and from kidneys removed at the time of renal failure due to the invasive nature and additional limitations of the currently available techniques. A non-invasive and direct method to assess the intrarenal microvasculature is needed to improve early detection and gauge the progression of microvascular alterations and monitor the success of therapeutic approaches.

Current imaging modalities, such as micro-computed tomography, magnetic resonance imaging, and contrast-enhanced ultrasound, have attempted to provide a non-invasive assessment of the intrarenal microvasculature in pre-clinical models of kidney diseases. However, each of these modalities has important limitations when translating into humans, including high cost, requiring long imaging times, using nephrotoxic contrast agents, radiation exposure, low spatial resolution, and poor reproducibility.

Super-resolution ultrasound (SRU) imaging is among the most rapidly advancing imaging techniques introduced to overcome the limitation of the inherent spatial resolution of ultrasound. With the use of non-nephrotoxic contrast microbubbles to break the diffraction limit of ultrasound, and the introduction of ultrasound localization microscopy which utilizes ultrafast frame rate imaging to reconstruct a super-resolved composite image, SRU has provided a paradigm-shifting tool for structural and functional evaluation of tissue microvasculature. However, in vivo, human imaging, and kidney imaging pose significant organ depth challenges (which results in ultrasound signals with lower signal-to-noise ratio) and physiologic and operator-induced motion (which reduces the available data accumulation time). Our team recently implemented advanced filtering and microbubble localization and tracking techniques to overcome these limitations, which extract only microbubble signals and reliably pinpoint the center of each microbubble from the extracted signals.

The investigators' broad objective is to deploy and evaluate the use of SRU imaging coupled with advanced post-processing techniques to assess the intrarenal microvasculature in patients with early ADPKD and healthy volunteers.

Participants in this study will have a renal ultrasound to determine intrarenal microvascular parameters, and an abdominal MRI to determine the patient's total kidney volume (TKV), and additional vascular parameters. In addition, participants will have a blood and a urine sample collected to determine biomarkers of endothelial function and injury.

ELIGIBILITY:
Inclusion Criteria (Patients with ADPKD):

* Male and female subjects 18 - 40 years of age, inclusive
* Previous diagnosis of ADPKD (based on Ravine et al. criteria)
* Class 1 according to imaging classification
* Estimated GFR> 90 mL/min/m2 (CKD-Epi equation)
* Ability to provide written, informed consent

Inclusion Criteria (Healthy Volunteers):

* Male and female subjects 18 - 40 years of age, inclusive
* Estimated GFR> 90 mL/min/m2 (CKD-Epi equation)
* Ability to provide written, informed consent

Exclusion Criteria (Patients with ADPKD):

* Class 2 according to imaging classification
* A concomitant systemic disease affecting the kidney (e.g., lupus, hepatitis B or C, amyloidosis)
* Diabetes mellitus (fasting glucose > 126 mg/dL or treatment with insulin or oral hypoglycemics).
* Predicted urine protein excretion in urinalysis >1 g/24 hrs.
* Subjects having contraindications to or interference with MRI assessments. [For example ferromagnetic metal prostheses, aneurysm clips, severe claustrophobia, large abdominal/back tattoos, etc.].
* History of hypersensitivity allergic reactions to ultrasound contrast agents
* High-risk cardiac disease (such as unstable hospital in-patients or ICU patients
* Patients that are part of an interventional study or are taking tolvaptan
* Female subjects that are pregnant

Exclusion Criteria (Healthy Volunteers):

* Family and/or personal history of kidney disease
* Concomitant systemic disease that may affect the kidney
* Diabetes mellitus
* Predicted urine protein excretion in >1 g/24 hrs, and or Abnormal urinalysis
* Pregnant or lactating women
* Subjects having contraindications to or interference with MRI assessments. [For example ferromagnetic metal prostheses, aneurysm clips, severe claustrophobia, large abdominal/back tattoos, etc.].
* History of hypersensitivity allergic reactions to ultrasound contrast agents
* High risk cardiac disease (such as unstable hospital in-patients or ICU patients

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with a previous diagnosis of ADPKD that meet the inclusion criteria, and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of intrarenal microvascular density in HV and patients with ADPKD | Baseline
  Renal vessel density as percentage, determined by SRU.
Assessment of intrarenal microvascular flow speed in HV and patients with ADPKD | Baseline
  Microvascular flow speed (mm/s), determined by SRU.
Assessment of intrarenal microvascular perfusion in HV and patients with ADPKD | Baseline
  Intrarenal perfusion (mm/s), determined by SRU.
Assessment of intrarenal tortuosity indices in HV and patients with ADPKD | Baseline
  Tortuosity indices defined as sum of angles metric (SOAM) (rad/mm), determined by SRU

SECONDARY OUTCOMES:
Inter-sonographer variability of the intrarenal microvasculature | Baseline
  Second US at the same visit performed by a different sonographer, and used to calculate the intraclass correlation coefficient
Day-to-day variability of intrarenal microvasculature in healthy volunteers | Baseline to 7 days
  A second US within 1-7 days is performed by the same sonographer, to determine the within-person variability for each of the primary outcome measures
Patient-to-patient variability in patients with ADPKD | Baseline
  Correlation between primary outcome measures and image class (A, B, C, D and E) as determined by the Image classification.

CONTACTS AND LOCATIONS:
Overall Officials: Maria V Irazabal, M.D., Ph.D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No